CLINICAL TRIAL: NCT00596583
Title: AQNA-DY001: A Double-Masked, Randomized Study of the Safety and Effectiveness of DYME as an Agent for Selective Staining of the Anterior Capsule During Cataract Surgery
Brief Title: DY001: Safety and Effectiveness of DYME as an Agent for Selective Staining of the Anterior Capsule During Cataract Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Aqumen Biopharmaceuticals, N.A. (Industry)
Responsible Party: Hardy Kagimoto, M.D. / C.E.O., Aqumen Biopharmaceuticals, N.A.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AQNA-DY001; US IND 75,735
Record Dates: First submitted 2008-01-09; First posted 2008-01-17 (Estimated); Last update posted 2009-03-02 (Estimated); Status verified 2009-02

CONDITIONS: Mature Cataracts

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- High Dose (Active Comparator)
  Interventions: Drug: DYME
- Low Dose (Active Comparator)
  Interventions: Drug: DYME

INTERVENTIONS:
Drug: DYME — 2ml of 0.25 mg/ml BBG 250 in sterile ophthalmic solution
  Arms: High Dose
Drug: DYME — 2ml of 0.05 mg/ml BBG 250 in sterile ophthalmic solution
  Arms: Low Dose

SUMMARY:
The primary objective of this study is to test the hypothesis that DYME is safe and effective as a drug to facilitate continuous curvilinear capsulorhexis (CCC) by selectively staining the anterior capsule. Secondary objectives are to compare the safety and effectiveness of DYME to that of a smaller dose of the same API.

ELIGIBILITY:
Inclusion Criteria:

* Have a cataract sufficiently opaque/mature/brunescent that, in the surgeon's assessment,a dye could facilitate surgery;
* Be aged at least 18 years old at the time of enrollment;
* Be able to tolerate a surgical procedure for up to 3 hours;
* Be in a medical condition suitable for cataract surgery;
* Able and willing to participate in study examinations and visit schedule; and
* Understand and freely consent to participate in the study.

Exclusion Criteria:

* In either eye, ocular infection or inflammation within the past 3 months;
* Known allergy to BBG 250;
* Uncontrolled intercurrent diseases including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, or cardiac arrhythmia;
* Active treatment for cancer or systemic infection within the past month;
* Active treatment with systemic corticosteroids within the past month;
* Previous participation in this Study for the contralateral eye;
* Participation in another clinical trial involving an investigational therapeutic during the past 30 days or 5.5 half-lives (if applicable), whichever is longer;
* Unwillingness to participate in the study or inability to give informed consent; or
* Any medical condition that in the opinion of the Investigator may compromise the research subject's safety or ability to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2007-04; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Optimal curvilinear capsulorrhexis with a single dose, as assessed by the surgeon based on the tissue dyed and subsequently removed. | During surgery
Uncomplicated discharge | one week post-op

SECONDARY OUTCOMES:
Quality of stain | during surgery
Intra-ocular safety of DYME as measured by best corrected visual acuity, corneal endothelial cell count, intraocular pressure, presence/absence of retained dye, duration of surgery, and the absence of dye related adverse events | 1-day and 1-week post-op

CONTACTS AND LOCATIONS:
Overall Officials: Hardy Kagimoto, M.D., Study Director — Aqumen Biopharmaceuticals, N.A.
Locations (21):
- United States (17):
  - McDonald Eye Associates, Fayetteville, Arkansas
  - Peace Laser Eye Center, Inglewood, California
  - Capitol City Surgery Center, Sacramento, California
  - The Eye Institute of West Florida, Largo, Florida
  - Center for Excellence in Eye Care, Miami, Florida
  - Eye Surgeons of Indiana, Indianapolis, Indiana
  - Silverstein Eye Centers, Kansas City, Missouri
  - St. John's Clinic Eye Specialists, Springfield, Missouri
  - Ballas Surgery Center, St Louis, Missouri
  - Wills Eye Surgery Center, Cherry Hill, New Jersey
  - Brar-Parekh Eye Associates, Woodland Park, New Jersey
  - Island Eye Surgicenter, Carle Place, New York
  - The Ohio State University Hospital, Columbus, Ohio
  - Eye Care Specialists, Kingston, Pennsylvania
  - Wills Eye Surgery Center, Philadelphia, Pennsylvania
  - Wills Surgery Center, Philadelphia, Pennsylvania
  - SMDV Surgery Center, Madison, Wisconsin
- India (4):
  - Narayana Nethralaya, Bangalore, Karnataka
  - Bhagwan Mahaveer Jain Hospital, Bangalore, Karnataka
  - The Mehta International Eye Institute & Colaba Eye Hospital, Mumbai, Maharashtra
  - Bombay City Eye Institute & Research Centre, Mumbai, Maharashtra